CLINICAL TRIAL: NCT02053376
Title: A Phase 2 Trial of Regorafenib as A Single Agent in Advanced and Metastatic Biliary Tract Carcinoma/Cholangiocarcinoma Patients Who Have Failed First-line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Bahary, MD (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Nathan Bahary, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-100
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Biliary Tract Carcinoma
Keywords: gallbladder cancer, biliary cancer, bile duct cancer, hepatobiliary cancer, Biliary Tract Carcinoma; Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Biliary Tract Neoplasms; Bile Duct Neoplasms; Cholangiocarcinoma | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- regorafenib (Experimental): Patients with advanced and metastatic biliary tract adenocarcinoma (cholangiocarcinoma) who had been treated with and failed first-line chemotherapy will be treated with regorafenib (120 mg) (160 mg for second and subsequent treatment cycles) orally once daily 21 days (3 weeks) on and 7 days (1 week) off in the 28-day (4-week) cycle
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — regorafenib (120 mg) (160 mg for second and subsequent treatment cycles)orally once daily 21 days (3 weeks) on and 7 days (1 week) off in the 28-day (4-week) cycle.
  Other Names: STIVARGA

SUMMARY:
Based on the facts of multiple pathways involvement in cholangiocarcinoma tumor genesis, including EGFR, Ras, Raf, VEGFR, and PDGFR, with evidence of overexpression of these proteins associated with tumor stage, prognosis and response to therapy. Multikinase inhibitor targeting multiple tumor pathways agent as regorafenib should be the ideal candidate for evaluating the anti-cancer activity for the disease as cholangiocarcinoma. More importantly, regorafenib likely holds promise in this disease setting with known effectiveness either as a single agent or in combination with cytotoxic chemotherapy agents in multiple solid tumors as above and the toxicity profile.

DETAILED DESCRIPTION:
Multiple pathways, including epidermal growth factor receptor (EGFR), Ras, Raf, Vascular Endothelial Growth Factor Receptors (VEGFR), and platelet-derived growth factor (PDGFR) appear to be involved in cholangiocarcinoma tumor genesis. Overexpression of these proteins has been shown to be associated with tumor stage, prognosis, and response to therapy. However, therapies targeting a single pathway have shown no clear benefit. A number of Phase 2 trials have been completed, or are underway, studying agents targeted to EGFR or VEGF - both as monotherapy and in combination with chemotherapy. These have shown varying increases in response rate, but have not found marked increases in progression-free or overall survival. This suggests that inhibition of multiple pathways simultaneously may be needed. Regorafenib, is an oral multikinase inhibitor targeting multiple tumor pathways, which has showed effectiveness as a single agent in multiple solid tumors.

Patients with advanced and metastatic biliary tract adenocarcinoma (cholangiocarcinoma) who had been treated with and failed first-line chemotherapy will be treated with regorafenib (120 mg) (160 mg for second and subsequent treatment cycles) orally once daily 21 days (3 weeks) on and 7 days (1 week) off in the 28-day (4-week) cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of biliary tract adenocarcinoma/cholangiocarcinoma (including primary intra- and extrahepatic diseases); pathologic confirmation may be from the primary or a metastatic site
* Must have locally advanced or distant metastatic disease that is not surgically curable
* Failed first-line chemotherapy (including systemic and local-regional therapy).
* Age ≥ 18 years.
* Life expectancy of at least ≥ 12 weeks (3 months).
* Performance status ECOG ≤ 1
* Adequate liver, kidney, and bone marrow function as assessed by the following laboratory requirements:

  * Total bilirubin ≤ 3.0 x the upper limit of normal (ULN) (biliary stenting or percutaneous biliary drainage are allowed for cancer related biliary obstruction)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5.0 x ULN
  * Alkaline phosphastase limit ≤ 2.5 x ULN (≤ 5.0 x ULN for subjects with intrahepatic involvement of their cancer)
  * Serum creatinine ≤ 1.5 x the ULN
  * International normalized ratio (INR)/partial thromboplastin time (PTT) ≤ 1.5 x ULN. (Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care).
  * Platelet count ≥ 75,000 /mm3
  * Hemoglobin (Hb) ≥ 9 g/dL,
  * Absolute neutrophil count (ANC) ≥ 1500/mm3.
  * Blood transfusion to meet the inclusion criteria will not be allowed.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Patients (men and women) of childbearing potential must agree to use Double Barrier method of birth control beginning at the signing of the ICF until at least 3 months after the last dose of study drug.
* Patients must be able to swallow and retain oral medication.
* Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.
* Uncontrolled hypertension (systolic pressure ≥140 mm Hg or diastolic pressure ≥ 90 mm Hg on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > Class II
  * Active coronary artery disease.
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Unstable angina (angina symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ Grade 3 within 4 weeks prior to prior to registration.
* Patients with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of the study registration.
* Previous exposure to Vascular endothelial growth factor (VEGF) inhibitor(s),
* Patients with any previously untreated or concurrent cancer that is distinct in primary site or histology from biliary tract cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Patients surviving a cancer that was curatively treated and without evidence of disease for more than 3 years prior to registration are allowed. All cancer treatments must be completed at least 3 years prior to prior to registration).
* Patients with phaeochromocytoma.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection > Grade 2.
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Renal failure requiring hemo-or peritoneal dialysis.
* Dehydration Grade ≥1
* Patients with seizure disorder requiring medication.
* Proteinuria ≥ Grade 3 (> 3.5 g/24 hours, measured by urine protein: creatinine ratio on a random urine sample).
* Active signs and symptoms of interstitial lung disease pleural effusion or ascites that causes respiratory compromise (≥ Grade 2 dyspnea).
* History of organ allograft (including corneal transplant).
* Known or suspected allergy or hypersensitivity to any of the study drug classes.
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment regorafenib. However, the palliative external beam radiation therapy (XRT) to non-targeted lesions is allowed.
* Prior use of regorafenib.
* Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 28 days prior to registration
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration (biliary stenting or percutaneous biliary drainage are not included).
* Use of any herbal remedy (e.g. St. John's Wort [Hypericum perforatum])

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01-07 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bahary, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Regorafenib: Patients with advanced and metastatic biliary tract adenocarcinoma (cholangiocarcinoma) who had been treated with and failed first-line chemotherapy will be treated with regorafenib (120 mg) (160 mg for second and subsequent treatment cycles) orally once daily 21 days (3 weeks) on and 7 days (1 week) off in the 28-day (4-week) cycle
  regorafenib: (120 mg) (160 mg for second and subsequent treatment cycles)orally once daily 21 days (3 weeks) on and 7 days (1 week) off in the 28-day (4-week) cycle.
Period: Overall Study
Arm/Group | Regorafenib
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who received at least one dose of regorafenib treatment.
Arm/Group | Regorafenib
Number analyzed (Participants) | 43
Age, Continuous [Mean (Full Range); unit: years] | 62.7 [34.5 to 82.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Duration of time from start of treatment to time of progression or death, whichever occurs first. Per RECIST version 1.1, Progressive Disease (PD) is defined as: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 4 years
Population: Patients who received at least one dose of regorafenib.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Regorafenib
Number analyzed (Participants) | 43
months | 3.58 [2.96 to 5.68]

2. Primary Outcome: Progression-free Survival (PFS) - Two or More Doses
Description: as for outcome 1
Time Frame: up to 4 years
Population: Patients who received two or more doses of regorafenib.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Regorafenib
Number analyzed (Participants) | 31
months | 3.91 [3.55 to 7.39]

3. Secondary Outcome: Proportion of Participants With Overall Response (OR)
Description: The number of patients who experienced a Partial Response (PR) + the number of patients who experienced a Complete Response (CR) / total number of response-evaluable patients. Per RECIST v1.1, Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 4 years
Population: Patients who received at least one dose of regorafenib and were evaluable for response
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 34
proportion of participants | 0.147 [0.060 to 0.285]

4. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of study treatment that patients remained alive.
Time Frame: Up to 4 years
Population: Patients who received at least one dose of regorafenib.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Regorafenib
Number analyzed (Participants) | 43
months | 5.55 [4.43 to 13.4]

5. Secondary Outcome: Overall Survival (OS) - Two or More Doses
Description: The length of time from the start of study treatment that patients remained alive.
Time Frame: Up to 4 years
Population: Patients who received two or more doses of regorafenib.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Regorafenib
Number analyzed (Participants) | 31
months | 9.43 [5.72 to 19.4]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: Number of patients who achieved Complete Response (CR) + number of patients who achieved Partial Response (PR) + number of patients who achieved Stable Disease (SD) / total number of response-evaluable patients. Per RECIST v1.1, Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study treatment.
Time Frame: Up to 4 years
Population: Patients who received at least one dose of regorafenib and were evaluable for response
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 34
proportion of participants | 0.706 [0.552 to 0.831]

7. Secondary Outcome: Changes in Cancer Antigen 19-9 (CA19-9) Level
Description: The difference between the levels of Cancer antigen 19-9 (CA19-9) prior to treatment compared to after treatment.
Time Frame: At baseline prior to treatment and after all treatment received, up to 4 years
Population: Patients who received at least one dose of regorafenib and for which CA19-9 levels were obtainable.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Regorafenib
Number analyzed (Participants) | 40
mg/dL
  Before Treatment | 100.6 [6.9 to 20558.0]
  After Treatment | 186.6 [8.0 to 28842.0]

8. Secondary Outcome: Change in Carcinoembryonic Antigen (CEA)
Description: The difference between the levels of Carcinoembryonic antigen (CEA) prior to treatment compared to after treatment. ng/ml
Time Frame: At baseline prior to treatment and after all treatment received, up to 4 years.
Population: Patients who received at least one dose of regorafenib.
Measure: Mean (90% Confidence Interval); unit: ng/ml
Arm/Group | Regorafenib
Number analyzed (Participants) | 35
ng/ml | 3.88 [1.11 to 6.90]

ADVERSE EVENTS:
Time Frame: Adverse event(s) data were collected over an approximately 4 year period of time.
Arm/Group | Regorafenib
All-Cause Mortality (participants affected / at risk) | 39/43
Serious Adverse Events (participants affected / at risk) | 27/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib (N=43)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 3
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 2
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Biliary tract infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Intracranial hemorrhage (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib (N=43)
Anemia (Blood and lymphatic system disorders) | 33
Sinus bradycardia (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 12
Flatulence (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 16
Chills (General disorders) | 5
Edema limbs (General disorders) | 6
Fever (General disorders) | 8
Pain (General disorders) | 13
General disorders and administration site conditions - Other, specify (General disorders) | 17
Fatigue (General disorders) | 31
Infections and infestations - Other, specify (Infections and infestations) | 4
Lymphocyte count increased (Investigations) | 3
INR increased (Investigations) | 5
Investigations - Other, specify (Investigations) | 5
Lipase increased (Investigations) | 6
Weight loss (Investigations) | 6
Neutrophil count decreased (Investigations) | 11
Creatinine increased (Investigations) | 12
Lymphocyte count decreased (Investigations) | 19
White blood cell decreased (Investigations) | 19
Blood bilirubin increased (Investigations) | 24
Alanine aminotransferase increased (Investigations) | 25
Alkaline phosphatase increased (Investigations) | 29
Platelet count decreased (Investigations) | 29
Aspartate aminotransferase increased (Investigations) | 33
Hyperglycemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 7
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 12
Hypernatremia (Metabolism and nutrition disorders) | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 18
Hyponatremia (Metabolism and nutrition disorders) | 28
Hypoalbuminemia (Metabolism and nutrition disorders) | 33
Hypophosphatemia (Metabolism and nutrition disorders) | 33
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Peripheral motor neuropathy (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 6
Urine discoloration (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 4
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 11
Hypotension (Vascular disorders) | 6
Hypertension (Vascular disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT02053376/Prot_SAP_000.pdf